CLINICAL TRIAL: NCT05336019
Title: Effectiveness of the Diabetes Self-management Coaching Program on the Clinical and Behavioral Parameters for Individuals With Type 2 Diabetes in the Ethiopian PC Setting: Mixed-methods Feasibility Randomized Controlled Trial
Brief Title: The Effect of a Diabetes Self-management Coaching Program for Type 2 Diabetes Patients in the Ethiopian PC.
Acronym: Primarycare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Fikadu Yehualashet, Mr., Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20224207
Record Dates: First submitted 2022-04-06; First posted 2022-04-20 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes; Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; self-management; Type 2 Diabetes; Coaching; Empowerment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Empowerment

STUDY DESIGN:
Intervention Model Description: A single-blinded, parallel-group feasibility Randomized Controlled Trial design.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked not be aware of the random assignment of study participants. Trained outcome assessors who are working in health facilities where participants are not selected will be recruited and involved in the data collection once either in baseline or end line evaluation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Diabetes self-management Coaching" (Experimental): A 12-week Diabetes self-management Coaching program and the usual care
  Interventions: Behavioral: Diabetes self-management Coaching
- "Usual Care" (Active Comparator): The control group will be assigned to 12 weeks usual care or routine diabetes service
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Diabetes self-management Coaching — A 12-week Diabetes self-management coaching program
  Other Names: Diabetes Health Coaching
  Arms: "Diabetes self-management Coaching"
Other: Usual care — Assigned to 12 weeks of usual care which includes a physical examination, history taking,, medication refill, lab investigation, and health education
  Other Names: routine service
  Arms: "Usual Care"

SUMMARY:
Background: Diabetes mellitus is the third most prevalent chronic disease globally. It is a metabolic disorder characterized by elevated blood glucose because of impaired insulin production, reduced insulin effectiveness, or both. It is a major contributor for physical disability and impaired quality of life. Diabetic Self-Management programs help to control blood glucose, reduce hospitalization, and increase compliance; however, the program is underutilized in the Primary Care settings globally; due to cognitive, financial, behavioral, and emotional factors. Health coaching is a client-centered self-management approach informed by behavioral change theories to empower individuals to identify their strengths and resources and achieve their health and wellness goals.

Purpose: The study's overarching goal is to determine whether implementing the Diabetes Self-Management (DSM) Coaching program can be effective and feasible for individuals with type diabetes in the Ethiopian primary care context.

Method: The study will employ a single-blinded feasibility randomized controlled trial followed by a concurrent mixed-method design. A block randomization technique with block size of 4 will be used to allocate eligible participants for the quantitative part. Structured outcome measures will be used to collect data on self-efficacy, self-care practice, and glycated hemoglobin A1c. Qualitative description approach with an in-depth interview method of data collection will be used to explore perspectives of participants, barriers and facilitators, and acceptability of the program. Mean, median and frequencies will be computed. Depending on the normality of the distribution and the number of participants, t-tests, x2 tests, sign tests, and ANOVA will be considered to analyze the data. Inductive qualitative content analysis approach will be followed to analyze qualitative data. Qualitative and quantitative data will be merged at result level for further interpretation and presented in discussion section.

Significance: The study will be used to determine the feasibility of the Diabetic Self-Management Coaching program in the Ethiopian primary care settings. Study participants will be benefited from the coaching program and will improve their self-efficacy, diabetes self-care practice, and blood glucose level. Furthermore, the study will have a paramount advantage to establish a foundation for future definitive trial that can prove effectiveness of the program.

DETAILED DESCRIPTION:
Primary Aim Objective 2. To determine the acceptability of implementing a DSM Coaching program in the Ethiopian PC setting.

The specific objectives are:

1.1. To assess the recruitment ability, adherence, retention ability, and satisfaction of the study participants.

1.2. To determine the fidelity of implementing the DSM Coaching program. Secondary Aim Objective 2. Evaluate the effectiveness of the DSM Coaching program on self-efficacy, self-care practice, and HbA1c among individuals with type 2 diabetes attending PC in Gondar town.

The specific objectives include- 2.1. To evaluate the effect of the DSM Coaching program on the self-efficacy of individuals with type 2 diabetes 2.2. To examine the effect of the DSM Coaching program on the self-care practice of individuals with type 2 diabetes.

2..3. To determine the effect of the DSM Coaching program on the HbA1C of individuals with type 2 diabetes.

Study participants assigned to intervention group will attend 12 weeks DSM Coaching program. This program has two components, four group based sessions and 4 individual home-based coaching. The control group will take the routine diabetes care for the same duration. The outcome will be assessed at baseline, after completing the intervention and after a two months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Attend diabetes care for at least 1 year
* Taking anti-diabetic medications
* Age between 18 -65 years
* HbA1c level >7% or Repeated FBS>130

Exclusion Criteria:

* Attend behavioral therapy program in the last 1 year
* Clinically confirmed mentally ill clients
* Pregnant
* Physically impaired (unable to see, hear, and walk)
* Clinically confirmed co-morbidity (Heart failure, cancer, stroke) which may interfere with their participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the DSM Coaching program | up to 1 year
  Acceptability measures the reaction of individual recipients-both study subjects and interventionists to the intervention(Bowen et al., 2009). It will be measured using a validated scale (B. J. Weiner et al., 2017). Mean scores will be used to categorize responses into acceptable and non-acceptable.
Recruitment rate | up to 1 year
  It is the proportion of eligible individuals willing to give consent and randomized to the study.
Ahernece rate | 1 year
  An intervention adherence is the participant's compliance with attending all group sessions, and all home-based coaching sessions.
Retention rate | 1year
  The ability of the program to retain participants in the study. The proportion of study participants who completed the study and evaluated at the end of the intervention T2 and end of follow-up T3.

SECONDARY OUTCOMES:
Diabetes self-efficacy | up to 1 year
  Diabetes self-efficacy will be measured using Stanford Self-Management Resource Center (SMRC) diabetes self-efficacy scale (SMRC, 2021). Mean scores will be computed to decide changes in values.
Diabetes self-care practice | up to 1 year
  The diabetes self-care practice will be measured using the Summary of Diabetes Self-Care Activity (SDSCA)(Toobert et al., 2000). Mean scores will be computed to decide changes in values.
Glycated Hemoglobin A1c (HbA1c) | up to 1 year
  HbA1c will be analyzed from a sample of whole blood using a chemistry machine at the University of Gondar hospital laboratory department. HbA1c < 7.0% is considered as the good glycemic control and HbA1c ≥ 7.0% will be considered as poorly controlled glucose level(Abera et al., 2022).

CONTACTS AND LOCATIONS:
Overall Officials: Fikadu A Yehualashet, Masters, Principal Investigator — Queen's University
Locations (1):
- Fikadu Ambaw Yehualashet, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
For the sake of confidentiality, participant data will not be shared. However, data will be disseminated in the form of publications, conference presentations, and local media. In addition, data may be shared on request.

REFERENCES:
- [Result] Alaofe H, Asaolu I, Ehiri J, Moretz H, Asuzu C, Balogun M, Abosede O, Ehiri J. Community Health Workers in Diabetes Prevention and Management in Developing Countries. Ann Glob Health. 2017 May-Aug;83(3-4):661-675. doi: 10.1016/j.aogh.2017.10.009. Epub 2017 Nov 22. PMID 29221543
- [Result] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Result] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Result] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness. JAMA. 2002 Oct 9;288(14):1775-9. doi: 10.1001/jama.288.14.1775. PMID 12365965
- [Result] Campos BM, Kieffer EC, Sinco B, Palmisano G, Spencer MS, Piatt GA. Effectiveness of a Community Health Worker-Led Diabetes Intervention among Older and Younger Latino Participants: Results from a Randomized Controlled Trial. Geriatrics (Basel). 2018 Sep;3(3):47. doi: 10.3390/geriatrics3030047. Epub 2018 Aug 2. PMID 30345345
- [Result] Chapman A, Browning CJ, Enticott JC, Yang H, Liu S, Zhang T, Thomas SA. Effect of a Health Coach Intervention for the Management of Individuals With Type 2 Diabetes Mellitus in China: A Pragmatic Cluster Randomized Controlled Trial. Front Public Health. 2018 Sep 19;6:252. doi: 10.3389/fpubh.2018.00252. eCollection 2018. PMID 30283767
- [Result] Chen RY, Huang LC, Su CT, Chang YT, Chu CL, Chang CL, Lin CL. Effectiveness of Short-Term Health Coaching on Diabetes Control and Self-Management Efficacy: A Quasi-Experimental Trial. Front Public Health. 2019 Oct 30;7:314. doi: 10.3389/fpubh.2019.00314. eCollection 2019. PMID 31737593
- [Result] Coleman CM, Bossick AS, Zhou Y, Hopkins-Johnson L, Otto MG, Nair AS, Willens DE, Wegienka GR. Introduction of a community health worker diabetes coach improved glycemic control in an urban primary care clinic. Prev Med Rep. 2020 Nov 27;21:101267. doi: 10.1016/j.pmedr.2020.101267. eCollection 2021 Mar. PMID 33364150
- [Result] Denneson, L. M., Ono, S. S., Trevino, A. Y., Kenyon, E., & Dobscha, S. K. (2020). The applicability of self-determination theory to health coaching: a qualitative analysis of patient experiences. Coaching: An International Journal of Theory, Research and Practice, 13(2), 163-175. https://doi.org/https://www.tandfonline.com/action/showCitFormats?doi=10.1080/17521882.2019.1673457
- [Result] Dineen-Griffin S, Garcia-Cardenas V, Williams K, Benrimoj SI. Helping patients help themselves: A systematic review of self-management support strategies in primary health care practice. PLoS One. 2019 Aug 1;14(8):e0220116. doi: 10.1371/journal.pone.0220116. eCollection 2019. PMID 31369582
- [Result] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Result] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Result] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Result] Engelhard C, Lonneman W, Warner D, Brown B. The implementation and evaluation of health professions students as health coaches within a diabetes self-management education program. Curr Pharm Teach Learn. 2018 Dec;10(12):1600-1608. doi: 10.1016/j.cptl.2018.08.018. Epub 2018 Sep 14. PMID 30527826
- [Result] Feleke BE, Feleke TE, Kassahun MB, Adane WG, Fentahun N, Girma A, Alebachew A, Misgan E, Desyibelew HD, Bayih MT, Seid O. Glycemic Control of Diabetes Mellitus Patients in Referral Hospitals of Amhara Region, Ethiopia: A Cross-Sectional Study. Biomed Res Int. 2021 Jan 16;2021:6691819. doi: 10.1155/2021/6691819. eCollection 2021. PMID 33532494
- [Result] Gearing RE, El-Bassel N, Ghesquiere A, Baldwin S, Gillies J, Ngeow E. Major ingredients of fidelity: a review and scientific guide to improving quality of intervention research implementation. Clin Psychol Rev. 2011 Feb;31(1):79-88. doi: 10.1016/j.cpr.2010.09.007. Epub 2010 Oct 7. PMID 21130938
- [Result] Glasgow RE, Davis CL, Funnell MM, Beck A. Implementing practical interventions to support chronic illness self-management. Jt Comm J Qual Saf. 2003 Nov;29(11):563-74. doi: 10.1016/s1549-3741(03)29067-5. PMID 14619349
- [Result] Gray KE, Hoerster KD, Taylor L, Krieger J, Nelson KM. Improvements in physical activity and some dietary behaviors in a community health worker-led diabetes self-management intervention for adults with low incomes: results from a randomized controlled trial. Transl Behav Med. 2021 Dec 14;11(12):2144-2154. doi: 10.1093/tbm/ibab113. PMID 34424331
- [Result] Gregg EW, Beckles GL, Williamson DF, Leveille SG, Langlois JA, Engelgau MM, Narayan KM. Diabetes and physical disability among older U.S. adults. Diabetes Care. 2000 Sep;23(9):1272-7. doi: 10.2337/diacare.23.9.1272. PMID 10977018
- [Result] Haas L, Maryniuk M, Beck J, Cox CE, Duker P, Edwards L, Fisher E, Hanson L, Kent D, Kolb L, McLaughlin S, Orzeck E, Piette JD, Rhinehart AS, Rothman R, Sklaroff S, Tomky D, Youssef G. National standards for diabetes self-management education and support. Diabetes Educ. 2012 Sep-Oct;38(5):619-29. doi: 10.1177/0145721712455997. No abstract available. PMID 22996411
- [Result] Hailu FB, Moen A, Hjortdahl P. Diabetes Self-Management Education (DSME) - Effect on Knowledge, Self-Care Behavior, and Self-Efficacy Among Type 2 Diabetes Patients in Ethiopia: A Controlled Clinical Trial. Diabetes Metab Syndr Obes. 2019 Nov 29;12:2489-2499. doi: 10.2147/DMSO.S223123. eCollection 2019. PMID 31819574
- [Result] Hayes E, McCahon C, Panahi MR, Hamre T, Pohlman K. Alliance not compliance: coaching strategies to improve type 2 diabetes outcomes. J Am Acad Nurse Pract. 2008 Mar;20(3):155-62. doi: 10.1111/j.1745-7599.2007.00297.x. PMID 18336692
- [Result] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Result] Jutterstrom L, Hornsten A, Sandstrom H, Stenlund H, Isaksson U. Nurse-led patient-centered self-management support improves HbA1c in patients with type 2 diabetes-A randomized study. Patient Educ Couns. 2016 Nov;99(11):1821-1829. doi: 10.1016/j.pec.2016.06.016. Epub 2016 Jun 17. PMID 27372525
- [Result] Kang M, Ragan BG, Park JH. Issues in outcomes research: an overview of randomization techniques for clinical trials. J Athl Train. 2008 Apr-Jun;43(2):215-21. doi: 10.4085/1062-6050-43.2.215. PMID 18345348
- [Result] Nigatu T. Epidemiology, complications and management of diabetes in Ethiopia: a systematic review. J Diabetes. 2012 Jun;4(2):174-80. doi: 10.1111/j.1753-0407.2011.00181.x. PMID 22212307
- [Result] Pamungkas RA, Chamroonsawasdi K. Self-management based coaching program to improve diabetes mellitus self-management practice and metabolic markers among uncontrolled type 2 diabetes mellitus in Indonesia: A quasi-experimental study. Diabetes Metab Syndr. 2020 Jan-Feb;14(1):53-61. doi: 10.1016/j.dsx.2019.12.002. Epub 2019 Dec 18. PMID 31887715
- [Result] Pirbaglou M, Katz J, Motamed M, Pludwinski S, Walker K, Ritvo P. Personal Health Coaching as a Type 2 Diabetes Mellitus Self-Management Strategy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Am J Health Promot. 2018 Sep;32(7):1613-1626. doi: 10.1177/0890117118758234. Epub 2018 Apr 15. PMID 29658286
- [Result] Raghupathi W, Raghupathi V. An Empirical Study of Chronic Diseases in the United States: A Visual Analytics Approach. Int J Environ Res Public Health. 2018 Mar 1;15(3):431. doi: 10.3390/ijerph15030431. PMID 29494555
- [Result] Resnick HE, Foster GL, Bardsley J, Ratner RE. Achievement of American Diabetes Association clinical practice recommendations among U.S. adults with diabetes, 1999-2002: the National Health and Nutrition Examination Survey. Diabetes Care. 2006 Mar;29(3):531-7. doi: 10.2337/diacare.29.03.06.dc05-1254. PMID 16505501
- [Result] Sherifali D. Diabetes coaching for individuals with type 2 diabetes: A state-of-the-science review and rationale for a coaching model. J Diabetes. 2017 Jun;9(6):547-554. doi: 10.1111/1753-0407.12528. Epub 2017 Feb 28. PMID 28084681
- [Result] Sherifali D, Jones H, Mullan Y. Diabetes self-management: what are we really talking about? Can J Diabetes. 2013 Feb;37(1):2-3. doi: 10.1016/j.jcjd.2013.01.003. Epub 2013 Mar 14. No abstract available. PMID 24070741
- [Result] Sherifali D, Viscardi V, Bai JW, Ali RM. Evaluating the Effect of a Diabetes Health Coach in Individuals with Type 2 Diabetes. Can J Diabetes. 2016 Feb;40(1):84-94. doi: 10.1016/j.jcjd.2015.10.006. PMID 26827684
- [Result] Siminerio LM, Piatt GA, Emerson S, Ruppert K, Saul M, Solano F, Stewart A, Zgibor JC. Deploying the chronic care model to implement and sustain diabetes self-management training programs. Diabetes Educ. 2006 Mar-Apr;32(2):253-60. doi: 10.1177/0145721706287156. PMID 16554429
- [Result] Smith LL, Lake NH, Simmons LA, Perlman A, Wroth S, Wolever RQ. Integrative Health Coach Training: A Model for Shifting the Paradigm Toward Patient-centricity and Meeting New National Prevention Goals. Glob Adv Health Med. 2013 May;2(3):66-74. doi: 10.7453/gahmj.2013.034. PMID 24416674
- [Result] Spieth PM, Kubasch AS, Penzlin AI, Illigens BM, Barlinn K, Siepmann T. Randomized controlled trials - a matter of design. Neuropsychiatr Dis Treat. 2016 Jun 10;12:1341-9. doi: 10.2147/NDT.S101938. eCollection 2016. PMID 27354804
- [Result] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Result] Wagner EH, Austin BT, Davis C, Hindmarsh M, Schaefer J, Bonomi A. Improving chronic illness care: translating evidence into action. Health Aff (Millwood). 2001 Nov-Dec;20(6):64-78. doi: 10.1377/hlthaff.20.6.64. PMID 11816692
- [Result] Wayne N, Perez DF, Kaplan DM, Ritvo P. Health Coaching Reduces HbA1c in Type 2 Diabetic Patients From a Lower-Socioeconomic Status Community: A Randomized Controlled Trial. J Med Internet Res. 2015 Oct 5;17(10):e224. doi: 10.2196/jmir.4871. PMID 26441467
- [Result] Werfalli M, Raubenheimer P, Engel M, Peer N, Kalula S, Kengne AP, Levitt NS. Effectiveness of community-based peer-led diabetes self-management programmes (COMP-DSMP) for improving clinical outcomes and quality of life of adults with diabetes in primary care settings in low and middle-income countries (LMIC): a systematic review and meta-analysis. BMJ Open. 2015 Jul 15;5(7):e007635. doi: 10.1136/bmjopen-2015-007635. PMID 26179646
- [Result] Werfalli MM, Kalula SZ, Manning K, Levitt NS. Does social support effect knowledge and diabetes self-management practices in older persons with Type 2 diabetes attending primary care clinics in Cape Town, South Africa? PLoS One. 2020 Mar 13;15(3):e0230173. doi: 10.1371/journal.pone.0230173. eCollection 2020. PMID 32168342
- [Result] Williams GC, McGregor HA, Zeldman A, Freedman ZR, Deci EL. Testing a self-determination theory process model for promoting glycemic control through diabetes self-management. Health Psychol. 2004 Jan;23(1):58-66. doi: 10.1037/0278-6133.23.1.58. PMID 14756604
- [Result] Wolever RQ, Simmons LA, Sforzo GA, Dill D, Kaye M, Bechard EM, Southard ME, Kennedy M, Vosloo J, Yang N. A Systematic Review of the Literature on Health and Wellness Coaching: Defining a Key Behavioral intervention in Healthcare. Glob Adv Health Med. 2013 Jul;2(4):38-57. doi: 10.7453/gahmj.2013.042. PMID 24416684
- [Result] Wong-Rieger D, Rieger FP. Health coaching in diabetes: empowering patients to self-manage. Can J Diabetes. 2013 Feb;37(1):41-4. doi: 10.1016/j.jcjd.2013.01.001. Epub 2013 Mar 14. PMID 24070747
- [Derived] Yehualashet FA, Kessler D, Bizuneh S, Donnelly C. Feasibility of diabetes self-management coaching program for individuals with type 2 diabetes in the Ethiopian primary care setting: a protocol for a feasibility mixed-methods parallel-group randomized controlled trial. Pilot Feasibility Stud. 2024 Apr 8;10(1):59. doi: 10.1186/s40814-024-01487-3. PMID 38589966